CLINICAL TRIAL: NCT06592547
Title: EFFECT of INTRAVENOUS METOPROLOL TARTRATE on MORTALITY in PATIENTS with SEPTIC SHOCK DUE to VENTILATOR-ASSOCIATED PNEUMONIA Thesis
Brief Title: Intravenous Metoprolol in Septic Shock
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Sherouk Rafik, Resident, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0106979
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Septic Shock; Ventilator Acquired Pneumonia
Keywords: Beta blockers; septic shock; Rate control; mortality
MeSH Terms: conditions — Shock, Septic; Pneumonia, Ventilator-Associated | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Metoprolol group (Active Comparator): The group that received intravenous metoprolol
  Interventions: Drug: Intravenous metoprolol tartrate
- Control group (Placebo Comparator): The group that received standard care
  Interventions: Other: Standard Care (in control arm)

INTERVENTIONS:
Drug: Intravenous metoprolol tartrate — An intravenous beta-blockers, recieved FDA approval
  Arms: Metoprolol group
Other: Standard Care (in control arm) — Standard care according to surviving sepsis campaign
  Arms: Control group

SUMMARY:
A RCT designed to assess the effect of giving intravenous beta-blockers in patients with septic shock after achieving hemodynamic stability. The principle of this study is to control heart rate allowing for better diastolic filling and thus better perfusion.

DETAILED DESCRIPTION:
A RCT, conducted at alexandria main university hospital, patients were divided into 2 groups, Control group which received the standard care for septic shock and metoprolol group which recieved intravenous metoprolol then patients were assessed for Blood pressure, heart rate, iv fluids needed, vasopressor doses and 28 days mortality

ELIGIBILITY:
Inclusion Criteria:

* The study population included adult patients (≥ 18 years) diagnosed with septic shock secondary to VAP with sinus tachycardia, from April 1, 2022, to April 31, 2023. Septic shock was defined according to the Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). VAP was identified as per the guidelines provided by the American Thoracic Society and Infectious Diseases Society of America.

Exclusion Criteria:

* Patients were excluded if they had contraindications to beta-blockers, had a history of heart failure, or had been receiving beta-blockers prior to the septic shock. Patients were also excluded if they developed complications from beta- blockers administration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
28-day Mortality | 28 days

SECONDARY OUTCOMES:
ICU stay | 28 days
ventilator days | 28 days
iv fluids | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Main university hospital, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided